CLINICAL TRIAL: NCT01075841
Title: A Korean Post-Marketing Surveillance Study On Erbitux (Cetuximab) In Patients With Recurrent And/Or Metastatic Squamous Cell Carcinoma Of The Head And Neck
Brief Title: A Post-marketing Surveillance Study on Erbitux in Combination With Platinum-based Chemotherapy in Metastatic/Recurrent Squamous Cell Cancer of the Head and Neck
Status: Withdrawn | Type: Observational
Why Stopped: After loss of orphan drug status in Korea, study was withdrawn due to Regulatory Authority request. Patients will be enrolled into NCT01075828 instead.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Head of Medical Department, Merck Serono Korea, an affiliate of Merck KGaA, Darmstadt, Germany
Other Study IDs: EMR 62241-510
Record Dates: First submitted 2010-02-24; First posted 2010-02-25 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2010-12

CONDITIONS: Neoplasms, Squamous Cell
Keywords: Head and neck neoplasms; Carcinoma, squamous cell; Cetuximab
MeSH Terms: conditions — Neoplasms, Squamous Cell; Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Cetuximab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cetuximab — Subjects who are eligible for Erbitux treatment according to the indication in the national label of Erbitux (i.e. where Erbitux is used in combination with platinum-based therapy for the treatment of subjects with recurrent and/or metastatic SCCHN) according to the approved national label as in routine clinical practice under the supervision of an investigator experienced in the use of antineoplastic medicinal products.
  Other Names: Erbitux

SUMMARY:
This is a prospective post-marketing surveillance (PMS) study to collect safety information from more than 600 subjects with recurrent and/or metastatic squamous cell cancer of the head and neck (SCCHN) treated with Erbitux as final evaluable cases. This PMS study is requested by the Korean Regulatory Authorities. After approval of new indication in Korea, there is a requirement to investigate more than 600 subjects during six years, to continue monitoring and provide further information about safety and toxicity in clinical practice.

DETAILED DESCRIPTION:
The PMS study is planned to be conducted within 6 years from the approval date of the new indication in approximately 50 institutions in Korea.

OBJECTIVES

Primary objective:

* To obtain safety information on the use of Erbitux in subjects with recurrent and/or metastatic SCCHN in terms of frequency and severity of adverse events (AEs)

Secondary objectives:

* To gather clinical efficacy information of the treatment

During the PMS period, each subject's background, subject's medical history (surgery, anti-cancer treatment), Erbitux treatment status, concurrent medication, response evaluation, status and reason of discontinuation, all AEs (regardless of the causal relationship to Erbitux), and abnormal results of laboratory tests will be collected. The PMS will be based on all cases treated with Erbitux at least once.

Erbitux will be prescribed to recurrent and/or metastatic SCCHN subjects according to the approved national label as in routine clinical practice under the supervision of an investigator experienced in the use of antineoplastic medicinal products. Prior to the first infusion, subjects will receive pre-medication with an antihistamine and a corticosteroid. The initial dose of Erbitux is 400 mg/m2 body surface area and the subsequent weekly doses are 250 mg/m2 each administered intravenously via in-line filtration with an infusion pump, gravity drip, or a syringe pump. The recommended infusion period for the initial dose is 120 minutes and for the subsequent weekly doses is 60 minutes with the maximum infusion rate not exceeding 10 mg/min, equivalent to 5 ml/min of Erbitux 2 mg/ml or 2ml/min of Erbitux 5mg/mL.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are eligible for Erbitux treatment according to the indication in the national label of Erbitux. The national label approved by Korea Food & Drug Administration is "Erbitux in combination with radiation therapy is indicated for the treatment of subjects with metastatic/recurrent SCCHN.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with recurrent and/or metastatic SCCHN undergoing treatment with Erbitux in Korea.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Safety | After approval of new indication till 6 years of PMS period
  Frequency and severity of all adverse events (AEs), regardless of the causal relationship to Erbitux

SECONDARY OUTCOMES:
Efficacy | Throughout 6 years of PMS period
  Best tumour response; time to progression; and duration of tumor response